CLINICAL TRIAL: NCT05081323
Title: Effectiveness of an Online Self-applied Psychological Treatment for Rat Phobia Guided by a Virtual Assistant in the Mexican Population: A Randomized Clinical Trial
Brief Title: Online Psychological Treatment for Rat Phobia Guided by a Virtual Assistant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Autonoma de Baja California (Other)
Collaborators: Universidad Internacional de Valencia (Other); Universidad Nacional Autonoma de Mexico (Other); Tecnológico Nacional de México (Unknown)
Responsible Party: Principal Investigator, María Victoria Meza Kubo, Principal Investigator, Universidad Autonoma de Baja California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 239
Record Dates: First submitted 2021-10-05; First posted 2021-10-18 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Specific Phobia; Anxiety Disorder
Keywords: Virtual therapeutic assistant; Small animal phobia; Exposure therapy; Self-applied treatment; Serious games; 360º videos
MeSH Terms: conditions — Phobia, Specific; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study has two arms, one is the experimental group that receives the treatment and the other is the comparison group that will receive treatment after the 2 months of the experimental group finished. The patients in both groups will be evaluated pre and post/treatment. The participants are assigned randomly to the intervention or comparison group.
Who Masked: Participant
Masking Description: The participants will not be aware the study includes two conditions. The conditions of the study are only known by the researchers and the Research Ethics Committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-applied treatment with THERA (Experimental): Participants in this group will use the Self-applied treatment with THERA for a maximum period of one month.
  Interventions: Behavioral: Self-applied treatment for phobias
- Control without treatment (No Intervention): Participants in this group keep on a waiting list, after one month, they will receive the self-applied treatment

INTERVENTIONS:
Behavioral: Self-applied treatment for phobias — The proposed treatment consists of four stages that use different visual elements to represent and replace a real rat in a gradual exposure treatment for specific phobia for animals. With the order of the stages, the intensity of the phobic stimulus increases. In each stage the participant is gradually exposed to a certain amount of elements that represent a phobic situation or object. Graduality considers an approach with realism, interaction, and intensity. The treatment also includes a virtual therapeutic assistant that guides, provides information, and tries to reduce any alteration captured by the participant's heart rate monitoring through deep breathing exercises.
  Arms: Self-applied treatment with THERA

SUMMARY:
The research work proposes an exposure treatment through a virtual therapeutic assistant called Thera, that interacts verbally with the patient, to guide and control exposure therapies for phobias to small animals delivered through several channels at the same time that it analyzes the Physiological records of the patient in real-time to determine their emotional state during the intervention.

In this study it is proposed to evaluate the efficacy of a self-applied treatment where the virtual assistant allows to gradually guide an exposure treatment for rat phobias, taking advantage of intelligent devices for patient monitoring and being considered to determine the progress of the treatment.

DETAILED DESCRIPTION:
Specific phobias are a common disorder that deteriorates the lives of people who suffer from them. Exposure therapies have been shown to reduce the symptoms produced. However, low- and middle-income countries have the lowest rate of treatment for specific phobia due to multiple barriers that prevent approaching mental health problems, such as the disparity between the number of people who need care and the availability of professionals who can provide psychological services. To reduce the gap in the treatment of mental health problems in low and middle-income countries, the use of internet-based interventions has been proposed since they reduce the cost, the availability of the service, the waiting time, and they can be guided by a minimum amount of therapeutic care, which allows a greater number of people to receive treatment. Among the most effective proposals that have emerged to carry out psychological interventions for Specific Phobia are self-applied treatments. However, one of the main challenges posed by self-administered interventions in reducing the dropout rate of participants, since it is difficult to engage participants, which leads to attrition and non-completion of treatment. Therefore, it is necessary to consider elements that are attractive and motivate the participants to engage with the treatment. One option to increase patient's adherence could be a virtual therapist assistant that is an application focused on the area of health therapies that uses interaction with the user based on voice commands, it requires a reduced cognitive learning load and are accessible to most of the people. The content of the intervention will be self-applied through a web application including the guidance of a virtual therapist assistant. In order to integrate the benefits that Internet-based interventions provides and the assistance of a virtual therapist to guide and personalize the progress of the treatment according to the user.

The study will have two groups : 1) experimental, where the participants carry out the self-applied treatment for rat phobia supported by the virtual therapist assistant; and 2) control, where participants are on a waiting list and afterwards receive the treatment.

The group assignment of participants will be randomized.

Participants in both groups will be measured pre and post the intervention. The measurements to be obtained are the following:

Fear scale. Anxiety scale. Sense of presence and judgment of reality. User's satisfaction. Perception of utility and ease of use. Patient improvement scale.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for specific phobia towards rats (with a mild to moderate symptomatology).
2. Have basic digital knowledge and skills (computer and internet use).
3. Have the necessary technological devices: email, computer / laptop, Smartphone, microphone, internet connection, and Bluetooth.
4. Sign the informed consent.

Exclusion Criteria:

1. Receiving another type of psychological or psychopharmacological treatment.
2. Being diagnosed with another type of anxiety disorder or some psychopathology.
3. Present any medical condition that puts the life of the person at risk (eg. heart disease, respiratory disease, pregnancy, among others).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change in the scores of the fear to the rats | From 2 to 4 weeks, depending on the development of the patient and the completion of the 4 sessions
  It is a questionnaire that has been adapted from the Fear of Spider Questionnaire for this, the word spiders have been modified for rats and the questions have been adapted to assess phobia rats. The Fear of Spiders Questionnaire has been adapted into Castilian Spanish, is a self-reported instrument that contains 18 items that assess fear of spiders. The items are answered on a seven-point Likert scale (0 = "it is not characteristic of me" up to 6 = "it is very characteristic of me"), the minimum score is 0 and the maximum score is 108. It is expected a statistically significant change (P < 0.05) for the fear of the rat.
Change on the avoidance of the presence of the rat. | From 2 to 4 weeks, depending on the development of the patient and the completion of the 4 sessions
  The Fear Questionnaire contains 23 items that evaluate a total of 5 subscales: agoraphobia, phobia of blood and wounds, social phobia, concern about feeling anxious and depressed as well as the assessment of the global present state of phobic symptoms. The first part contains 16 items that assess the frequency with which a person avoids phobic situations on a scale of 0 to 8 (0 = I do not avoid it and 8 = I always avoid it), the minimum score is 0 and the maximum score is 120 and the second part contains 7 items that evaluate: 1) the degree to which you are worried about feeling anxious and depressed (0 = almost nothing and 8 = very severely worried), the minimum score is 0 and the maximum is 40; 2) the overall severity of the phobic symptoms (0 = there is no phobia and 8 = very severely disturbing /disabling), the minimum score is 0 and the maximum score is 8. It is expected a statistically significant change (P < 0.05) for the avoidance and fear of the presence of the rat.
Change in anxiety symptoms | From 2 to 4 weeks, depending on the development of the patient and the completion of the 4 sessions
  The State-Trait Anxiety Inventory will be used. It contains 40 statements that are grouped into two self-assessment scales that measure two different dimensions of anxiety, contain four response options with different criteria for each dimension: 1) Anxiety-trait (almost never, some sometimes, frequently and almost always); 2) Anxiety-state (no, little, regular and a lot). Answers are scored 1, 2, 3, and 4 in the positive reagents (the higher the score, the higher anxiety) and 4, 3, 2, and 1 in negative items (the higher the score, the lower the anxiety). The score can range from a minimum score of 20, up to a maximum score of 80. It is expected a statistically significant change (P < 0.05) for symptoms of anxiety.

SECONDARY OUTCOMES:
Level of satisfaction with self-administered treatment with a virtual assistant | From 2 to 4 weeks, depending on the development of the patient and the completion of the 4 sessions
  The Client Satisfaction Questionnaire contains 8 questions with a total score ranging from 8 to 32 that measures the level of satisfaction of the self-administered treatment with an assistant virtual Thera; and contains a question that explores the degree to which the treatment is perceived as aversive, it is measured on a scale from 0 (not at all) to 10 (very much).
Perception of the level of effectiveness and ease of use of the self-applied system for fear of rats with a virtual assistant | From 2 to 4 weeks, depending on the development of the patient and the completion of the 4 sessions
  The Telehealth Usability Questionnaire will be used, it contains 12 questions with 7 response options (1 = disagree and 7 = agree) that evaluate the participant's perception in relation to the effectiveness and ease of use of the self-administered treatment.
Degree of presence and degree of Judgment of reality | From 2 to 4 weeks, depending on the development of the patient and the completion of the 4 sessions
  Two questions will be used that uses a Likert scale from 0 to 10 (0 = not at all and 10 = too much), the first question assesses the degree to which the patient feels immersed in the virtual environment; the second assesses the degree to which the patient perceives the virtual experience as real (exposure of the rats through 360 ° videos).
Patient perception in the change of fear of rats. | From 2 to 4 weeks, depending on the development of the patient and the completion of the 4 sessions
  An item adapted from the Clinical Global Impression scale will be used, the question assesses the perception that the patient has in relation to the change in fear of rats after treatment. The question contains a 7-point scale (1 = much better and 7 = much worse). The minimum score is 0 and the maximum score is 7.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia M. González Lozoya, MD, Study Chair — UNIVERSIDAD AUTONOMA DEL ESTADO DE BAJA CALIFORNIA

IPD SHARING:
Plan to Share IPD: Yes
The information will be available in a private server or in a server of the journal(s) that we will publish the articles that will be the result of this study.
Supporting Information: ICF
Time Frame: This data will be available approximately in April 2023 and it will be permanently available. It will be shared in the databases of the journal where the article(s) will be published.
Access Criteria: Through the servers of the journal(s) where we will publish the articles.

REFERENCES:
- [Background] Albor YC, Benjet C, Mendez E, Medina-Mora ME. Persistence of Specific Phobia From Adolescence to Early Adulthood: Longitudinal Follow-Up of the Mexican Adolescent Mental Health Survey. J Clin Psychiatry. 2017 Mar;78(3):340-346. doi: 10.4088/JCP.15m10569. PMID 28394508
- [Background] Campos D, Breton-Lopez J, Botella C, Mira A, Castilla D, Mor S, Banos R, Quero S. Efficacy of an internet-based exposure treatment for flying phobia (NO-FEAR Airlines) with and without therapist guidance: a randomized controlled trial. BMC Psychiatry. 2019 Mar 6;19(1):86. doi: 10.1186/s12888-019-2060-4. PMID 30841930
- [Background] Felix IB, Guerreiro MP, Cavaco A, Claudio AP, Mendes A, Balsa J, Carmo MB, Pimenta N, Henriques A. Development of a Complex Intervention to Improve Adherence to Antidiabetic Medication in Older People Using an Anthropomorphic Virtual Assistant Software. Front Pharmacol. 2019 Jun 21;10:680. doi: 10.3389/fphar.2019.00680. eCollection 2019. PMID 31281256
- [Background] Jimenez-Molina A, Franco P, Martinez V, Martinez P, Rojas G, Araya R. Internet-Based Interventions for the Prevention and Treatment of Mental Disorders in Latin America: A Scoping Review. Front Psychiatry. 2019 Sep 13;10:664. doi: 10.3389/fpsyt.2019.00664. eCollection 2019. PMID 31572242
- [Background] Wechsler TF, Kumpers F, Muhlberger A. Inferiority or Even Superiority of Virtual Reality Exposure Therapy in Phobias?-A Systematic Review and Quantitative Meta-Analysis on Randomized Controlled Trials Specifically Comparing the Efficacy of Virtual Reality Exposure to Gold Standard in vivo Exposure in Agoraphobia, Specific Phobia, and Social Phobia. Front Psychol. 2019 Sep 10;10:1758. doi: 10.3389/fpsyg.2019.01758. eCollection 2019. PMID 31551840
- [Background] Brown TA, Di Nardo PA & Barlow DH. Anxiety Disorders Interview Schedule for DSM-IV (ADIS-IV): Client Interview Schedule. Oxford University Press. 1994.
- [Background] Morán AL, Ramírez-Fernández C & Meza-Kubo V. Design of smart objects of fear with a taxonomy of factors affecting the user experience of exposure therapy systems for small-animal phobias. Journal of Ambient Intelligence and Humanized Computing. 2020
- [Result] Bibiloni N, Torre AC, Angles MV, Terrasa SA, Vazquez Pena FR, Sommer J, Plazzotta F, Luna D, Mazzuoccolo LD. [Validation of a Spanish questionnaire on telemedicine usability]. Medicina (B Aires). 2020;80(6):649-653. Spanish. PMID 33254109
- [Result] Hemyari C, Dolatshahi B, Sahraian A, Koohi-Hosseinabadi O, Zomorodian K. Evaluation of the Effectiveness of One- and Multi-Session Exposure-Based Treatments in Reducing Biological and Psychological Responses to Rat Phobia Among Students. Psychol Res Behav Manag. 2020 Aug 12;13:665-679. doi: 10.2147/PRBM.S256781. eCollection 2020. PMID 32848483
- [Result] Juan MC, Alcaniz M, Monserrat C, Botella C, Banos RM, Guerrero B. Using augmented reality to treat phobias. IEEE Comput Graph Appl. 2005 Nov-Dec;25(6):31-7. doi: 10.1109/mcg.2005.143. No abstract available. PMID 16315475
- [Result] Marks IM, Mathews AM. Brief standard self-rating for phobic patients. Behav Res Ther. 1979;17(3):263-7. doi: 10.1016/0005-7967(79)90041-x. No abstract available. PMID 526242
- [Result] Palma-Gomez A, Herrero R, Banos R, Garcia-Palacios A, Castaneiras C, Fernandez GL, Llull DM, Torres LC, Barranco LA, Cardenas-Gomez L, Botella C. Efficacy of a self-applied online program to promote resilience and coping skills in university students in four Spanish-speaking countries: study protocol for a randomized controlled trial. BMC Psychiatry. 2020 Apr 5;20(1):148. doi: 10.1186/s12888-020-02536-w. PMID 32248795
- [Result] Ruiz-Garcia A, Valero-Aguayo L. Multimedia intervention for specific phobias: A clinical and experimental study. Psicothema. 2020 Aug;32(3):298-306. doi: 10.7334/psicothema2020.87. PMID 32711663
- [Result] Díaz-Guerrero R, & Spielberger CD. IDARE: Inventario de ansiedad: rasgo-estado. El Manual Moderno. 1975.
- [Result] Guy W. ECDEU Assessment Manual for Psychopharmacology. Rockville, MD: US Department of Heath, Education, and Welfare Public Health Service Alcohol, Drug Abuse, and Mental Health Administration. 1976.
- [Derived] Gonzalez-Lozoya SM, Meza-Kubo V, Dominguez-Rodriguez A, Ramirez-Fernandez C, Bautista-Valerio E, Moreyra-Jimenez L, Moran AL. An internet-based self-applied rat phobia treatment using a Virtual Therapy Assistant: Study protocol for a randomized controlled trial. PLoS One. 2023 Feb 15;18(2):e0281338. doi: 10.1371/journal.pone.0281338. eCollection 2023. PMID 36791089

DOCUMENTS (1):
  • Informed Consent Form (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/23/NCT05081323/ICF_001.pdf